CLINICAL TRIAL: NCT05841485
Title: A Comparative Analysis of Coronary Microvascular Dysfunction in Stable Angina Patients With and Without Severe COVID-19 History
Brief Title: COVID-19 Microvascular Evaluation Trial
Acronym: COMET-19
Status: Recruiting | Type: Observational
Sponsor: Lithuanian University of Health Sciences (Other)
Collaborators: Klaipėda University (Other)
Responsible Party: Principal Investigator, Ali Aldujeli, Cardiovascular disease consultant, Lithuanian University of Health Sciences
Other Study IDs: LUHSKC- 301
Record Dates: First submitted 2023-04-30; First posted 2023-05-03 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: COVID-19; Coronary Microvascular Dysfunction
Keywords: Coronary Microvascular Dysfunction; Stable angina; COVID-19; Mechanical ventilation; Coronary flow reserve; Index of microvascular resistance
MeSH Terms: conditions — COVID-19; Angina, Stable

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Stable angina patients with a history of severe COVID-19 infection requiring mechanical ventilation: Patients with a history of severe COVID-19 infection (confirmed by a polymerase chain reaction test) requiring mechanical ventilation. This group includes patients who have been recently diagnosed with stable angina and have previously experienced a severe COVID-19 infection that necessitated mechanical ventilation support during their illness.
  Interventions: Diagnostic Test: Assessment of coronary microvascular dysfunction using intracoronary pressure-temperature wire
- Patients with stable angina without a history of COVID-19 (Group B): Patients without a history of COVID-19. This group consists of patients who have been diagnosed with stable angina but have no history of COVID-19 infection. This group serves as a comparison group to assess the potential impact of severe COVID-19 infection on coronary microvascular dysfunction in patients with stable angina.
  Interventions: Diagnostic Test: Assessment of coronary microvascular dysfunction using intracoronary pressure-temperature wire

INTERVENTIONS:
Diagnostic Test: Assessment of coronary microvascular dysfunction using intracoronary pressure-temperature wire — The primary assessment method in this study is the measurement of coronary microvascular dysfunction using a pressure-temperature wire to determine coronary flow reserve (CFR) and index of microvascular resistance (IMR).

SUMMARY:
The COMET trial is an observational, cross-sectional study aimed at comparing the incidence of coronary microvascular dysfunction (CMD) in patients with stable angina who have a history of severe COVID-19 infection requiring mechanical ventilation (Group A) to those without a history of COVID-19 (Group B). A total of 102 participants will be recruited, with 51 patients in each group.

Data will be collected on participants' demographic information, medical history, and COVID-19 infection history (confirmed by PCR test). CMD measurement will be performed using a pressure-temperature wire to assess the coronary flow reserve and index of microcirculatory resistance. In addition, information on participants' current medications will be gathered. The study will employ statistical analysis tools to compare CMD incidence between the two groups and assess the impact of various factors such as age and sex on CMD incidence. The results of the COMET trial will provide valuable insights into the effects of severe COVID-19 infection on CMD in patients with stable angina.

DETAILED DESCRIPTION:
The COMET trial is an observational, cross-sectional study that aims to compare the incidence of coronary microvascular dysfunction (CMD) in patients with stable angina who have a history of severe COVID-19 infection requiring mechanical ventilation (Group A) to those without a history of COVID-19 (Group B). A total of 102 participants will be recruited, with 28 patients in each group.

The study will be conducted at two university hospitals: Seamen's Branch, Department of Cardiology, Klaipeda University Hospital, Klaipeda, Lithuania, and the Hospital of Lithuanian University of Health Sciences Kaunas clinics, Kaunas, Lithuania. The anticipated study duration is 6 months.

CMD measurement will involve assessing coronary flow reserve (CFR), fractional flow reserve (FFR), and index of microvascular resistance (IMR) using the CoroFlow system (Coroventis Research AB, Uppsala, Sweden). After diagnostic coronary angiography is performed and no significant visible lesion is identified, nitroglycerin will be administered through the intracoronary catheter. A calibrated coronary physiology wire (Pressure Wire X; Abbott Vascular, Santa Clara, CA, USA) will be equalized to the guide catheter pressure at the sinus of the aorta and advanced to the distal two-thirds of the left anterior descending artery. Three milliliters of normal saline will be administered through the guiding catheter in triplicates during rest and during maximal hyperemia, which will be induced by injecting intracoronary adenosine.

Data analysis will be performed using appropriate statistical tests, such as the chi-squared test or Fisher's exact test for categorical data and the independent-samples t-test or Mann-Whitney U test for continuous data, as appropriate. Multivariable regression analysis will be used to assess the impact of various factors, such as age and sex, on CMD incidence.

The primary outcome measure for this study will be the incidence of CMD in both groups, as measured by both coronary flow reserve (CFR) and index of microvascular resistance (IMR) using the pressure-temperature wire. A potential secondary outcome measure could be the relationship between CMD severity and the severity of the patients' COVID-19 infection.

Safety monitoring and adverse event reporting procedures will be in place to ensure patient safety. All adverse events occurring during the study will be recorded and reported to the appropriate institutional review boards and regulatory authorities. Serious adverse events will be reported to the principal investigator within 24 hours of the study team's awareness of the event. The study team will regularly review adverse event data to assess patient safety and make any necessary modifications to the study protocol.

The results of the COMET trial will provide valuable insights into the effects of severe COVID-19 infection on CMD in patients with stable angina.

ELIGIBILITY:
Here's a detailed outline of the eligibility criteria, including inclusion, exclusion, and withdrawal criteria for the COMET trial. Please review and let me know if you need any further clarification or have additional information to provide.

Inclusion Criteria:

1. Patients with a clinical diagnosis of stable angina, consulted by a cardiovascular consultant and referred to undergo diagnostic coronary angiography.
2. Patients who are able to provide informed consent.
3. For Group A: Patients with a history of severe COVID-19 infection requiring mechanical ventilation, confirmed by a PCR test.
4. For Group B: Patients without a history of COVID-19 infection.

Exclusion Criteria:

1. Patients with unstable angina or acute coronary syndrome.
2. Patients with a history of myocardial infarction, percutaneous coronary intervention, or coronary artery bypass graft surgery.
3. Patients with known structural heart disease or valvular heart disease.
4. Patients who are unable to undergo intracoronary pressure-temperature wire measurement of CMD due to contraindications or other medical reasons.

Withdrawal Criteria:

1. Withdrawal of informed consent by the participant at any time during the study.
2. Development of an unstable medical condition or complication that prevents the participant from completing the study or makes it unsafe for them to continue.
3. Identification of exclusion criteria after enrollment that should have precluded the participant's inclusion in the study.
4. Non-compliance with study procedures or protocol deviations that may affect the validity of the study results.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population for the COMET trial consists of adult patients (aged 40 -80 years) with a clinical diagnosis of stable angina.
  The study population will be divided into two groups:
  Group A: Patients with a history of severe COVID-19 infection requiring mechanical ventilation, confirmed by a polymerase chain reaction test. This group represents individuals with stable angina who have experienced a severe COVID-19 infection and later on developed stable angina symptoms.
  Group B: Patients without a history of COVID-19 infection. This group serves as a comparison group to assess the potential differences in CMD incidence among patients with stable angina who have not been affected by COVID-19 infection.
Sampling Method: Non-Probability Sample
Enrollment: 102 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of coronary microvascular dysfunction | up to 1 month
  Incidence of coronary microvascular dysfunction in both groups, as measured by both coronary flow reserve (CFR) and index of microvascular resistance (IMR) using the pressure-temperature wire.

CONTACTS AND LOCATIONS:
Locations (1):
- Lithuanian University of Health Sciences, Kaunas, Lithuania

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Tsai TY, Aldujeli A, Haq A, Murphy P, Unikas R, Zaliaduonyte-Peksiene D, Braukyliene R, Kiernan TJ, Revaiah PC, Miyashita K, Tobe A, Oshima A, Celeutkiene J, Sharif F, Garg S, Tatarunas V, Onuma Y, Serruys PW. Diagnostic performance of exercise stress testing findings and coronary microvascular dysfunction in patients with angina with non-obstructive coronary artery disease. Heart. 2025 Aug 27:heartjnl-2025-325769. doi: 10.1136/heartjnl-2025-325769. Online ahead of print. PMID 40866120
- [Derived] Aldujeli A, Tsai TY, Haq A, Puipaite K, Braukyliene R, Tatarunas V, Zaliaduonyte D, Unikas R, Renkens M, Revaiah PC, Miyashita K, Tobe A, Oshima A, Sharif F, Lesauskaite V, Spertus JA, Garg S, Onuma Y, Brilakis ES, Serruys PW. Impact of severe COVID-19 infection on coronary microvascular dysfunction in ANOCA patients: A cross-sectional study. Atherosclerosis. 2025 Aug;407:120389. doi: 10.1016/j.atherosclerosis.2025.120389. Epub 2025 Jun 2. PMID 40483738

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-01): https://cdn.clinicaltrials.gov/large-docs/85/NCT05841485/Prot_SAP_000.pdf